CLINICAL TRIAL: NCT05561907
Title: Enteral Anastomosis for the Treatment of Gastric Outlet Obstruction: A Randomized Controlled Study Comparing Endoscopic Versus Surgical Gastrojejunostomy
Acronym: EAT-GO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Petros Benias, Director of Endoscopic Surgery, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1130
Record Dates: First submitted 2022-09-13; First posted 2022-09-30 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Gastric Outlet Obstruction
Keywords: Gastric outlet obstruction; GOO; Periampullary malignancy; Periampullary cancer; Surgical gastrojejunostomy; Endoscopic gastrojejunostomy; Gastrojejunostomy; Enteral anastamosis
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1 ratio to surgical gastrojejunostomy (SGJ) or endoscopic gastrojejunostomy (EGJ).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical gastrojejunostomy (SGJ) (Active Comparator): An anastomosis will be created between the stomach and the proximal loop of the jejunum during a laparoscopic surgical procedure.
  Interventions: Procedure: Surgical gastrojejunostomy (SGJ)
- Endoscopic gastrojejunostomy (EGJ) (Experimental): A stent is placed between the stomach and adjacent small intestine under endoscopic ultrasound guidance during an upper endoscopic procedure.
  Interventions: Procedure: Endoscopic gastrojejunostomy (EGJ)

INTERVENTIONS:
Procedure: Surgical gastrojejunostomy (SGJ) — Laparoscopic gastrojejunostomy
  Arms: Surgical gastrojejunostomy (SGJ)
Procedure: Endoscopic gastrojejunostomy (EGJ) — Endoscopic ultrasound (EUS) guided gastrojejunostomy
  Arms: Endoscopic gastrojejunostomy (EGJ)

SUMMARY:
Gastric outlet obstruction (GOO) occurs commonly in malignancies involving the periampullary region (cancers originating in the head of the pancreas, duodenum, bile duct, or ampulla) or the distal stomach. GOO not only causes debilitating symptoms such as nausea, vomiting, inability to tolerate oral intake, and prevents adequate nutritional intake. Therefore, providing therapy for GOO is imperative to improve the quality of life, and nutritional status of these patients, as well as allow them to continue receiving their cancer treatment

DETAILED DESCRIPTION:
After potential subjects are screened from the physicians' schedules, they will be assessed for further inclusion criteria. They will be presented with the informed consent form for their review. Once they have been given the opportunity to review and ask questions, they will sign the consent form and from this point will be considered enrolled into the study.

After signing the informed consent, subjects will be randomized to one of the two cohorts in a 1:1 manner.

On the day of their assigned procedures, subjects will be asked several quality of life questionnaires to obtain a baseline status.

Data will be collected during and immediately following the procedure to assess for any possible adverse events.

Follow-up data will be completed at the following timepoints: 1-day, 2-day, 3-day, 4-day, and 7-day, 30-day, 3-month, 6-month, and 1-year post-procedure.

QOL Scoring Systems GOOSS- Gastric Outlet Obstruction Symptom Score

* 1 Inadequate or no oral intake
* 2 Liquids/thickened liquids
* 3 Semisolids/ low residue
* 4 unmodified

GFS- Gut Function Score from Lowe et al 2002

* 0 Profuse vomiting
* 1 Nausea and occasional vomiting
* 2 Nausea only
* 3 Normal gut function

Pre-Procedure Variables to Record Demographic

* Gender
* Weight
* BMI
* Cancer Type

Clinical Parameters

* GOOSS
* Gut Function Score
* Karnofsky Performance Scale

Procedural Parameters

* EUS-GJ: presence of ascites, able to pass scope beyond obstruction, use of wire to stabilize position, Length of procedure, intraprocedural AEs, Stent size used, successful completion of procedure
* Laparoscopic GJ: presence of ascites, length of procedure, intraprocedural AEs, conversion to open GJ, successful completion of procedure

Post-procedure Hospitalization Daily Function

* GOOSS
* Gut Function Score
* Time to initiation of oral intake liquids
* Time to initiation of oral intake solids
* Time to discharge
* Post procedural AEs

  30 Day Outcomes
* GOOSS
* Gut Function Score
* Karnofsky Performance Scale
* Weight/BMI
* Able to tolerate TB approved chemotherapeutic regimen

ELIGIBILITY:
Inclusion Criteria:

1. Periampullary malignancy (pancreas, bile duct, ampulla, duodenum) extending to the distal duodenum (D3) or distal (antrum) gastric cancer
2. Symptoms of gastric outlet obstruction (at least 2 of 4 required):

   1. post prandial vomiting,
   2. abdominal pain,
   3. inability to tolerate PO,
   4. imaging consistent with GOO
3. Gastric Outlet Obstruction Scoring System (GOOSS) Score of 0 (no oral intake) or 1 (liquids only)
4. Age >18 years old
5. Life expectancy greater than 2 months or failed duodenal stenting
6. Surgical Candidate/Tolerate General Anesthesia
7. Unresectable or metastatic disease

Exclusion Criteria:

1. Age< 18 years old
2. Pregnancy
3. Intestinal obstruction distal to the Ligament of Treitz
4. Evidence of other luminal strictures of the GI tract
5. Previous gastric or periampullary surgery
6. Inability to complete quality of life surveys (QOLS)
7. Presence of abdominal ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of solid oral intake without symptoms of GOO | 1 year
  Days to initiation of solid oral intake will be measured from randomization to first day of intake of soft solid foods, as indicated by a GOOSS score of 2

SECONDARY OUTCOMES:
Safety of procedure | 1 year
  All adverse events (AEs) occurring after treatment will be graded according to ASGE lexicon. A subject will be considered to have had an adverse event if they had one or more adverse events, and they will be considered to have had a serious adverse event (SAE) if they had one or more serious adverse events
Technical success of procedure | 1 year
  Technical success is defined as adequate deployment and positioning of the stent(s) for EGJ or technical possibility to create an anastomosis for SGJ.
Clinical success of procedure | 1 year
  Clinical success is defined as improvement to a GOOSS score of 2 or 3 (oral intake of soft solid foods or resumption of full diet) without additional intervention.
Time to discharge | 1 year
  Length of stay will be measured from randomization to discharge alive. All patients will be followed until discharge. Patients who die in hospital will be considered censored and time from randomization to death will be used.
Change in BMI | 3 months
  BMI will be measured immediately prior to the procedure, and at one month and three months after the procedure.
Change in albumin levels | 3 months
  Albumin levels will be measured immediately prior to the procedure, and at one month and three months after the procedure.
Change in Gastric Outlet Obstruction Symptom Score (GOOSS) | 1 year
  The Gastric Outlet Obstruction Symptom Score (GOOSS) scale is as follows, whereas a score of 1 is the worst and a score of 4 is the best:
  1. Inadequate or no oral intake
  2. Liquids/thickened liquids
  3. Semisolids/ low residue
  4. Unmodified
  GOOSS will be recorded at each of the following timepoints:
  * immediately prior to the procedure
  * immediately post-procedure
  * 1-day post-procedure
  * 2-days post-procedure
  * 3-days post-procedure
  * 4-days post-procedure
  * 7-days post-procedure,
  * 30-days post-procedure
  * 3-months post-procedure
  * 6-months post-procedure
  * 1-year post-procedure
Change in Gut Function Score (GFS) | 1 year
  Gut Function Score (GFS) scale is as follows, whereas a score of 1 is the worst and a score of 3 is the best:
  0. Profuse vomiting
  1. Nausea and occasional vomiting
  2. Nausea only
  3. Normal gut function
  GFS will be recorded at each of the following timepoints:
  * Immediately prior to the procedure
  * Immediately post-procedure
  * 1-day post-procedure
  * 2-days post-procedure
  * 3-days post-procedure
  * 4-days post-procedure
  * 7-days post-procedure,
  * 30-days post-procedure
  * 3-months post-procedure
  * 6-months post-procedure
  * 1-year post-procedure
Karnofsky Performance Scale (KPS) | 30 Days
  Karnofsky Performance Scale is measured on a scale of 0 to 100 as follows, with a score of 0 being the worst and a score of 100 being the best:
  100 - Normal; no complaints; no evidence of disease. 90 - Able to carry on normal activity; minor signs or symptoms of disease. 80 - Normal activity with effort; some signs or symptoms of disease. 70 - Cares for self; unable to carry on normal activity or to do active work. 60 - Requires occasional assistance, but is able to care for most of their personal needs.
  50 - Requires considerable assistance and frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospital admission is indicated although death not imminent.
  20 - Very sick; hospital admission necessary; active supportive treatment necessary.
  10 - Moribund; fatal processes progressing rapidly. 0 - Dead
  KPS will be recorded pre-procedure and at 30-days post-procedure.
Chemotherapeutic regimen tolerance | 30 Days
  Ability to tolerate TB approved chemotherapeutic regimen

CONTACTS AND LOCATIONS:
Overall Officials: Petros Benias, MD, Principal Investigator — Northwell Health; Arvind Trindade, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorusso D, Giliberti A, Bianco M, Lantone G, Leandro G. Stomach-partitioning gastrojejunostomy is better than conventional gastrojejunostomy in palliative care of gastric outlet obstruction for gastric or pancreatic cancer: a meta-analysis. J Gastrointest Oncol. 2019 Apr;10(2):283-291. doi: 10.21037/jgo.2018.10.10. PMID 31032096
- [Background] Troncone E, Fugazza A, Cappello A, Del Vecchio Blanco G, Monteleone G, Repici A, Teoh AYB, Anderloni A. Malignant gastric outlet obstruction: Which is the best therapeutic option? World J Gastroenterol. 2020 Apr 28;26(16):1847-1860. doi: 10.3748/wjg.v26.i16.1847. PMID 32390697
- [Background] Maetani I, Inoue H, Sato M, Ohashi S, Igarashi Y, Sakai Y. Peroral insertion techniques of self-expanding metal stents for malignant gastric outlet and duodenal stenoses. Gastrointest Endosc. 1996 Oct;44(4):468-71. doi: 10.1016/s0016-5107(96)70102-5. PMID 8905371
- [Background] Tonozuka R, Tsuchiya T, Mukai S, Nagakawa Y, Itoi T. Endoscopic Ultrasonography-Guided Gastroenterostomy Techniques for Treatment of Malignant Gastric Outlet Obstruction. Clin Endosc. 2020 Sep;53(5):510-518. doi: 10.5946/ce.2020.151. Epub 2020 Sep 23. PMID 32962331
- [Background] Khashab M, Alawad AS, Shin EJ, Kim K, Bourdel N, Singh VK, Lennon AM, Hutfless S, Sharaiha RZ, Amateau S, Okolo PI, Makary MA, Wolfgang C, Canto MI, Kalloo AN. Enteral stenting versus gastrojejunostomy for palliation of malignant gastric outlet obstruction. Surg Endosc. 2013 Jun;27(6):2068-75. doi: 10.1007/s00464-012-2712-7. Epub 2013 Jan 9. PMID 23299137
- [Background] Jeurnink SM, Steyerberg EW, van Hooft JE, van Eijck CH, Schwartz MP, Vleggaar FP, Kuipers EJ, Siersema PD; Dutch SUSTENT Study Group. Surgical gastrojejunostomy or endoscopic stent placement for the palliation of malignant gastric outlet obstruction (SUSTENT study): a multicenter randomized trial. Gastrointest Endosc. 2010 Mar;71(3):490-9. doi: 10.1016/j.gie.2009.09.042. Epub 2009 Dec 8. PMID 20003966
- [Background] Jeurnink SM, Steyerberg EW, Hof Gv, van Eijck CH, Kuipers EJ, Siersema PD. Gastrojejunostomy versus stent placement in patients with malignant gastric outlet obstruction: a comparison in 95 patients. J Surg Oncol. 2007 Oct 1;96(5):389-96. doi: 10.1002/jso.20828. PMID 17474082
- [Background] Itoi T, Itokawa F, Uraoka T, Gotoda T, Horii J, Goto O, Moriyasu F, Moon JH, Kitagawa Y, Yahagi N. Novel EUS-guided gastrojejunostomy technique using a new double-balloon enteric tube and lumen-apposing metal stent (with videos). Gastrointest Endosc. 2013 Dec;78(6):934-939. doi: 10.1016/j.gie.2013.09.025. PMID 24237949
- [Background] Khashab MA, Kumbhari V, Grimm IS, Ngamruengphong S, Aguila G, El Zein M, Kalloo AN, Baron TH. EUS-guided gastroenterostomy: the first U.S. clinical experience (with video). Gastrointest Endosc. 2015 Nov;82(5):932-8. doi: 10.1016/j.gie.2015.06.017. Epub 2015 Jul 26. PMID 26215646
- [Background] Khashab MA, Tieu AH, Azola A, Ngamruengphong S, El Zein MH, Kumbhari V. EUS-guided gastrojejunostomy for management of complete gastric outlet obstruction. Gastrointest Endosc. 2015 Oct;82(4):745. doi: 10.1016/j.gie.2015.05.017. Epub 2015 Jun 16. No abstract available. PMID 26092615
- [Background] Carbajo AY, Kahaleh M, Tyberg A. Clinical Review of EUS-guided Gastroenterostomy (EUS-GE). J Clin Gastroenterol. 2020 Jan;54(1):1-7. doi: 10.1097/MCG.0000000000001262. PMID 31567785
- [Background] Barthet M, Binmoeller KF, Vanbiervliet G, Gonzalez JM, Baron TH, Berdah S. Natural orifice transluminal endoscopic surgery gastroenterostomy with a biflanged lumen-apposing stent: first clinical experience (with videos). Gastrointest Endosc. 2015 Jan;81(1):215-8. doi: 10.1016/j.gie.2014.09.039. PMID 25527056
- [Background] Ge PS, Young JY, Dong W, Thompson CC. EUS-guided gastroenterostomy versus enteral stent placement for palliation of malignant gastric outlet obstruction. Surg Endosc. 2019 Oct;33(10):3404-3411. doi: 10.1007/s00464-018-06636-3. Epub 2019 Feb 6. PMID 30725254
- [Background] Kerdsirichairat T, Irani S, Yang J, Brewer Gutierrez OI, Moran R, Sanaei O, Dbouk M, Kumbhari V, Singh VK, Kalloo AN, Khashab MA. Durability and long-term outcomes of direct EUS-guided gastroenterostomy using lumen-apposing metal stents for gastric outlet obstruction. Endosc Int Open. 2019 Feb;7(2):E144-E150. doi: 10.1055/a-0799-9939. Epub 2019 Jan 30. PMID 30705945
- [Background] James TW, Greenberg S, Grimm IS, Baron TH. EUS-guided gastroenteric anastomosis as a bridge to definitive treatment in benign gastric outlet obstruction. Gastrointest Endosc. 2020 Mar;91(3):537-542. doi: 10.1016/j.gie.2019.11.017. Epub 2019 Nov 20. PMID 31759034
- [Background] Wannhoff A, Ruh N, Meier B, Riecken B, Caca K. Endoscopic gastrointestinal anastomoses with lumen-apposing metal stents: predictors of technical success. Surg Endosc. 2021 May;35(5):1997-2004. doi: 10.1007/s00464-020-07594-5. Epub 2020 May 1. PMID 32358692
- [Background] Itoi T, Ishii K, Ikeuchi N, Sofuni A, Gotoda T, Moriyasu F, Dhir V, Teoh AY, Binmoeller KF. Prospective evaluation of endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy bypass (EPASS) for malignant gastric outlet obstruction. Gut. 2016 Feb;65(2):193-5. doi: 10.1136/gutjnl-2015-310348. Epub 2015 Aug 17. No abstract available. PMID 26282674
- [Background] Tyberg A, Perez-Miranda M, Sanchez-Ocana R, Penas I, de la Serna C, Shah J, Binmoeller K, Gaidhane M, Grimm I, Baron T, Kahaleh M. Endoscopic ultrasound-guided gastrojejunostomy with a lumen-apposing metal stent: a multicenter, international experience. Endosc Int Open. 2016 Mar;4(3):E276-81. doi: 10.1055/s-0042-101789. PMID 27004243
- [Background] Khashab MA, Bukhari M, Baron TH, Nieto J, El Zein M, Chen YI, Chavez YH, Ngamruengphong S, Alawad AS, Kumbhari V, Itoi T. International multicenter comparative trial of endoscopic ultrasonography-guided gastroenterostomy versus surgical gastrojejunostomy for the treatment of malignant gastric outlet obstruction. Endosc Int Open. 2017 Apr;5(4):E275-E281. doi: 10.1055/s-0043-101695. PMID 28382326
- [Background] Perez-Miranda M, Tyberg A, Poletto D, Toscano E, Gaidhane M, Desai AP, Kumta NA, Fayad L, Nieto J, Barthet M, Shah R, Brauer BC, Sharaiha RZ, Kahaleh M. EUS-guided Gastrojejunostomy Versus Laparoscopic Gastrojejunostomy: An International Collaborative Study. J Clin Gastroenterol. 2017 Nov/Dec;51(10):896-899. doi: 10.1097/MCG.0000000000000887. PMID 28697151
- [Background] Brewer Gutierrez OI, Nieto J, Irani S, James T, Pieratti Bueno R, Chen YI, Bukhari M, Sanaei O, Kumbhari V, Singh VK, Ngamruengphong S, Baron TH, Khashab MA. Double endoscopic bypass for gastric outlet obstruction and biliary obstruction. Endosc Int Open. 2017 Sep;5(9):E893-E899. doi: 10.1055/s-0043-115386. Epub 2017 Sep 13. PMID 28924596
- [Background] Chen YI, Itoi T, Baron TH, Nieto J, Haito-Chavez Y, Grimm IS, Ismail A, Ngamruengphong S, Bukhari M, Hajiyeva G, Alawad AS, Kumbhari V, Khashab MA. EUS-guided gastroenterostomy is comparable to enteral stenting with fewer re-interventions in malignant gastric outlet obstruction. Surg Endosc. 2017 Jul;31(7):2946-2952. doi: 10.1007/s00464-016-5311-1. Epub 2016 Nov 10. PMID 27834024
- [Background] Chen YI, James TW, Agarwal A, Baron TH, Itoi T, Kunda R, Nieto J, Bukhari M, Gutierrez OB, Sanaei O, Moran R, Fayad L, Khashab MA. EUS-guided gastroenterostomy in management of benign gastric outlet obstruction. Endosc Int Open. 2018 Mar;6(3):E363-E368. doi: 10.1055/s-0043-123468. Epub 2018 Mar 7. PMID 29527559
- [Background] Chen YI, Kunda R, Storm AC, Aridi HD, Thompson CC, Nieto J, James T, Irani S, Bukhari M, Gutierrez OB, Agarwal A, Fayad L, Moran R, Alammar N, Sanaei O, Canto MI, Singh VK, Baron TH, Khashab MA. EUS-guided gastroenterostomy: a multicenter study comparing the direct and balloon-assisted techniques. Gastrointest Endosc. 2018 May;87(5):1215-1221. doi: 10.1016/j.gie.2017.07.030. Epub 2017 Jul 24. PMID 28750837
- [Background] Antonelli G, Kovacevic B, Karstensen JG, Kalaitzakis E, Vanella G, Hassan C, Vilmann P. Endoscopic ultrasound-guided gastro-enteric anastomosis: A systematic review and meta-analysis. Dig Liver Dis. 2020 Nov;52(11):1294-1301. doi: 10.1016/j.dld.2020.04.021. Epub 2020 Jun 3. PMID 32505567
- [Background] Fan W, Tan S, Wang J, Wang C, Xu H, Zhang L, Liu L, Fan Z, Tang X. Clinical outcomes of endoscopic ultrasound-guided gastroenterostomy for gastric outlet obstruction: a systematic review and meta-analysis. Minim Invasive Ther Allied Technol. 2022 Feb;31(2):159-167. doi: 10.1080/13645706.2020.1792500. Epub 2020 Jul 16. PMID 32672479